CLINICAL TRIAL: NCT04612114
Title: Ring-type Pulse Oximeter for Evaluation for Sleep Assessment Study (ROSA Study)
Brief Title: Pulse Oximeter for Sleep Evaluation
Acronym: ROSA
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Belun Technology Company Limited (Other)
Responsible Party: Principal Investigator, Makoto Kawai, Clinical Associate Professor, Stanford University
Other Study IDs: 53979
Record Dates: First submitted 2020-10-22; First posted 2020-11-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; pulse oximeter; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Possible OSA: Patients with OSA symptoms (snoring, excessive daytime sleepiness or witnessed apnea, etc.)
  Interventions: Diagnostic Test: Belun Ring

INTERVENTIONS:
Diagnostic Test: Belun Ring — Simultaneous recording of Belun Ring data (pulse oximeter, pulse rate and actigraphy) and standard of care PSG will be performed for one night.

SUMMARY:
The investigators will conduct this study to validate Belun Ring for sleep assessment. The investigators will compare Belun Ring data collection and overnight in-lab polysomnography (PSG) measures of SDB and sleep architecture in adults with OSA symptoms.

The investigators propose to recruit a total of 40 participants with symptoms of obstructive sleep apnea. The investigators will i) validate the overall accuracy, sensitivity and specificity of Belun Ring to assess SDB and sleep architecture, using PSG analysis as a gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 80 years old. Ideally balanced for sex and age (18 to 80 years old)

   * No more than 75% of subjects in one bin of: (male, female)
   * No more than 50% of subjects in one age-group (18-29, 30-39, 40-49, 50-59, 60-80)
2. Patients with OSA symptoms (snoring, excessive daytime sleepiness or witnessed apnea, etc.)
3. Without any unstable medical or psychiatric co-morbidities that would be expected to interfere with the study.
4. If taking any medication, must be on a stable dose of medication for a month
5. Able to read and understand English

Exclusion Criteria:

1. Presence of any significant systemic or unstable medical condition which could lead to difficulty complying with the protocol, suicidality, current regular use of psychiatric medications, opiates, or thyroid medications, dementia, current substance abuse, post-traumatic or psychotic disorders, bipolar disorder; any significant neurologic disease, including possible and probable dementia, Parkinson's or Huntington's disease, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of significant head trauma, history of alcohol or substance use disorder within the past 2 years (DSM V criteria);
2. If positive airway pressure (PAP) titration study or split night study (diagnostic and PAP titration study combined)
3. Under 18 or over 80 years of age

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: i) 40 participants ii) All enrollment will be at Stanford iii) Patients with obstructive sleep apnea will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Validation with gold-standard polysomnography (PSG) recording | through study completion, an average of 1 year
  Concordance rate of respiratory disturbance index (RDI) from Belun Ring and apnea-hypopnea Index (AHI) from PSG

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Kawai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No